CLINICAL TRIAL: NCT00060892
Title: A Phase II Double-Blind, Randomized, Placebo-Controlled Study to Assess the Safety and Efficacy of AMG0001 to Improve Perfusion in Critical Leg Ischemia
Brief Title: Study of HGF Via Plasmid Vector to Improve Perfusion in Critical Limb Ischemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AnGes USA, Inc. (Industry)
Responsible Party: Prannath Marrott, M.D., AnGes Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG-CLI-0202
Record Dates: First submitted 2003-05-15; First posted 2003-05-16 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Arterial Occlusive Disease; Peripheral Vascular Disease; Ischemia
Keywords: Critical Limb Ischemia
MeSH Terms: conditions — Arterial Occlusive Diseases; Peripheral Vascular Diseases; Ischemia; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): 0.4 mg AMG0001 on days 0, 14, and 28
  Interventions: Genetic: HGF plasmid
- 2 (Active Comparator): 4.0 mg AMG0001 on days 0, 14, and 28
  Interventions: Genetic: HGF plasmid
- 3 (Active Comparator): 4.0 mg AMG0001 on days 0 and 28; placebo on day 14
  Interventions: Genetic: HGF plasmid
- 4 (Placebo Comparator): Placebo (saline) on days 0, 14, and 28
  Interventions: Genetic: HGF plasmid

INTERVENTIONS:
Genetic: HGF plasmid — Intramuscular injections into index leg on Days 0, 14, and 28

SUMMARY:
The primary purpose of this study was to assess the overall safety of different dose regimens of AMG0001 (HGF transferred via plasmid vector) as well as evaluate the improvement of blood perfusion in subjects with critical limb ischemia (CLI). This study also evaluated the improvement in wound healing without adverse effects on the quality of life, as well as the potential reduction of amputation, mortality and rest pain in the CLI population.

DETAILED DESCRIPTION:
The primary goal of this study was to assess the safety of AMG0001, detect potential angiogenesis response to AMG0001 treatment and to correlate these changes to clinical endpoints dependent upon improvement in tissue perfusion for relief of CLI complications. The objectives of this study were to:

* Assess the overall safety of different exposure regimens of AMG0001 in the CLI subject population.
* Evaluate the potential effect of angiogenesis associated with different doses and dose regimens of AMG0001 as measured by improvement in tissue perfusion.
* Evaluate the activity of different exposure regimens of AMG0001 to benefit clinical outcomes of reduction of amputation and mortality, wound healing, rest-pain reduction and improvement in subject's ability to function without adverse consequences on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have one or more clinical indications diagnostic of CLI such as: distal extremity pain at rest that requires the subject to use analgesics for >2 weeks; or peripheral ischemic ulcer(s); or areas of gangrene.
* The subject will have a TcPO2 of </= 40 mmHg.
* Subjects will have one or both of the following hemodynamic indicators of severe peripheral arterial occlusive disease: (a) Ankle systolic pressure of </= 70 mmHg; (b)Toe systolic pressure </= 50 mmHg.
* The subject is a poor candidate for standard revascularization treatment options for peripheral arterial disease, based on inadequate bypass conduit, unfavorable anatomy, or poor operative risk.
* Subject has signed an informed consent form either directly or through a legally authorized representative
* If female, the subject must be (a) at least one year post-menopausal, or (b) surgically sterile, or (c) if the subject is of child-bearing potential, she must have been practicing contraception for at least 12 weeks prior to entering the study.
* If subject is of reproductive potential, he or she must be using an accepted and effective (barrier) form of birth control during the study.
* Subjects will be on a statin and an anti-platelet agent as part of their standard of care and must be stable on these regimens for at least 4 weeks prior to treatment.

Exclusion Criteria:

* Subjects, who in the opinion of the investigator, have a vascular disease prognosis that indicates they would require a major amputation (at or above the ankle) within 4 weeks of start of treatment.
* Subjects with a diagnosis of Buerger's disease (Thromboangitis Obliterans).
* Subjects with hemodynamically significant aorto-iliac occlusive disease.
* Subjects who have had a revascularization procedure within 12 weeks prior to treatment initiation that remains patent. Revascularization procedures that are evidenced to have failed for >2 weeks prior to treatment initiation are acceptable.
* Subjects who require a change in their hypertension medication as part of their standard of care within 4 weeks prior to treatment.
* Evidence or history of malignant neoplasm (clinical, laboratory or imaging), except for basal cell carcinoma of the skin.
* Subjects who have proliferative diabetic retinopathy or severe, non-proliferative retinopathy
* Subjects with end stage renal disease (ESRD) defined as significant renal dysfunction evidenced by a creatinine of > 2.5, or receiving chronic hemodialysis therapy.
* A subject who has hepatic cirrhosis, viral hepatitis, or is HIV positive.
* Subjects with a clinically significant liver enzyme abnormality (i.e., AST or ALT more than two times the upper limit of normal and/or bilirubin more than 50% the upper limit of normal).
* Subjects requiring the use of hyperbaric oxygen treatment for wound healing during the screening and 6 month follow-up period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2003-04; Primary Completion 2006-05 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Tissue perfusion as measured by TcPO2 | 6 months

SECONDARY OUTCOMES:
Ulcer healing | 6 months

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Cardiology, P.C., Birmingham, Alabama
  - Central Arkansas Veteran's Healthcare System, Little Rock, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Falk Cardiovascular Research Center, Stanford, California
  - VA Medical Center Surgical Service (112), Washington D.C., District of Columbia
  - Basptist Hospital, Pensacola, Florida
  - University of South Florida College of Medicine, Tampa, Florida
  - American Cardiovascular Research Institute, Atlanta, Georgia
  - University of Chicago Hospitals, Chicago, Illinois
  - The Care Group, LLC, Indianapolis, Indiana
  - The Ochsner Heart and Vascular Institute, Metairie, Louisiana
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Dartmouth - Hitchcock Medical Center, Lebanon, New Hampshire
  - Diabetes Foot and Ankle Center, New York, New York
  - NYPH-NY Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Jobst Vascular Center, Toledo, Ohio
  - Medical College of Ohio, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Baylor College of Medicine, Houston, Texas
  - Peripheral Vascular Associates, San Antonio, Texas

REFERENCES:
- [Derived] Powell RJ, Simons M, Mendelsohn FO, Daniel G, Henry TD, Koga M, Morishita R, Annex BH. Results of a double-blind, placebo-controlled study to assess the safety of intramuscular injection of hepatocyte growth factor plasmid to improve limb perfusion in patients with critical limb ischemia. Circulation. 2008 Jul 1;118(1):58-65. doi: 10.1161/CIRCULATIONAHA.107.727347. Epub 2008 Jun 16. PMID 18559703